CLINICAL TRIAL: NCT06580158
Title: The Clinical Utility of Artificial Intelligence-enabled Electrocardiograms in the Outpatient Practice - Diagnosing Aortic Stenosis and Diastolic Dysfunction
Brief Title: AI in Outpatient Practice for Diagnosing Aortic Stenosis and Diastolic Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jae K. Oh, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 24-000100
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Aortic Stenosis; Diastolic Dysfunction
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients who are completing an outpatient electrocardiogram (ECG) at the Mayo Clinic.
  Interventions: Device: AI-ECG Dashboard; Diagnostic Test: Point of care ultrasound (POCUS)

INTERVENTIONS:
Device: AI-ECG Dashboard — Patients standard of care ECG's will be processed through the AI-ECG Dashboard
Diagnostic Test: Point of care ultrasound (POCUS) — Patients will undergo a ultrasound to confirm diagnosis of atrial stenosis or diastolic dysfunction.

SUMMARY:
Two recently developed artificial intelligence-enabled electrocardiogram (AI-ECG) models have been developed to detect aortic stenosis (AS) and diastolic dysfunction (DD). AI-ECG for AS has a sensitivity of 78% and specificity of 74%, and AI-ECG for DD has a sensitivity of 83% and specificity of 80%. However, these models have never been prospectively applied to diagnose AS or DD, which may be useful for patients and providers from a diagnostic and prognostic perspective and especially in settings where access to higher- level medical care is limited. In this study, we aim to determine the clinical utility of these AI-ECG models by prospectively applying them to an outpatient cohort and then completing a focused point-of-care ultrasound to evaluate those who are AI-ECG positive for AS and DD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age must have a clinical scheduled ECG performed.

Exclusion Criteria:

* < 59 years of age
* Is not scheduled for a clinical ECG
* Unable to provide consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are completing an outpatient electrocardiogram (ECG) at the Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive AI-ECG | Baseline
  Positive AI-ECG will be determined by the sensitivity, specificity, positive predictive value, and negative predictive value.
Number of studies with reasonable image quality in patients with positive AI-ECG | Baseline
  Image quality will be determined by sonographers at the time of imaging and will be scored on a scale from 1-4:
  1. Excellent , sufficient for publication
  2. Good, sufficient for data analysis
  3. Fair, just enough for data analysis without complete views
  4. Poor, not usable for data analysis

SECONDARY OUTCOMES:
Number of times the AI ECG and TTE (transthoracic echocardiogram) are statistically comparative | Baseline
  Will be compared using parametric (2-sample t-test) and non-parametric tests (Wilcoxon rank sum test) for continuous variables, and the χ2 test or Fisher exact test for nominal variables. A p-value of < 0.05 will be categorized as significant for the statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jae Oh, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No